CLINICAL TRIAL: NCT07121361
Title: Evaluation of the Efficacy of a Mouthwash Formulation for Minor Oral Ulcers: A Triple-Blind Randomized Controlled Trial
Brief Title: Effectiveness of Recurrent Aphthous Stomatitis Mouthwash System for the Treatment of Oral Ulcers
Acronym: RASMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: G. d'Annunzio University (Other)
Responsible Party: Principal Investigator, Felice Lorusso, Senior Researcher, Department of Innovative Technologies in Medicine and Dentistry, University "G.d'Annunzio" of Chieti-Pescara, G. d'Annunzio University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RA/0362820; RA/0362820 (Other: Territorial Ethics Committee of the Abruzzi Region, Italy (C.Et.R.A.) ))
Record Dates: First submitted 2025-08-01; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Aphthous Ulcer; Recurrent Aphthous Stomatitis
Keywords: Ulcers; Oral Hygiene; Oral care
MeSH Terms: conditions — Stomatitis, Aphthous; Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DNA mouthwash (Active Comparator): The compound is characterized by a formulation that ensures effective action on the film-forming component. The presence of DNA fractions increases the viscosity of the solutions and increases the hydration of the mucous membranes with a consequent improvement in trophism for oral ulcers.
  The treatment indications are to delay and prevent oral ulcers and the formation of bacterial plaque; prevent irritation of the gums and oral cavity, even in wearers of prostheses and orthodontic implants accompanied by problems with dental support structures; after tooth extraction; before and after any dental surgery. The patients will be instructed to rinse the mouth and ulcers with the mouthwash twice a day after oral hygiene for 14 days
  Interventions: Device: Mouthwash Product
- Placebo mouthwash (Placebo Comparator): The placebo will be deprived by all components. The patients will be instructed to rinse the mouth and ulcers with the mouthwash twice a day after oral hygiene for 14 days
  Interventions: Device: Control

INTERVENTIONS:
Device: Mouthwash Product — DNA mouthwash
  Arms: DNA mouthwash
Device: Control — Placebo mouthwash
  Arms: Placebo mouthwash

SUMMARY:
The purpose of the present research is to evaluate the efficacy of a gel formulation for a total treatment of 14 days for the treatment of traumatic or aphthous oral ulcers.

DETAILED DESCRIPTION:
Primary Objective

Evaluation of the clinical efficacy of the treatment using the following scores and clinical parameters:

Pain intensity, measured using the VAS (Visual Analogue Scale), consisting of a 10 cm line, where 0 indicates no pain and 10 indicates intense pain.

Size of each ulcer.

Secondary Objectives

Evaluation of the following scores and clinical parameters:

1. Registration of the superficial temperature of the mucous membranes using Infrared Thermography.
2. Ulcer Severity Score (USS).

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one well-defined oral ulcer.
* Patients with no cognitive disorders able to provide mouthwash treatment independently

Exclusion Criteria:

* Proven intolerance or allergy to the product.
* Patients with a hematological deficit such as anemia, iron deficiency, vitamin B12 and/or folic acid
* No systemic diseases including ulcerative colitis, Crohn's disease, Behçet's syndrome with recurrent aphthous lesions; alcohol and tobacco consumption;
* No history of allergies;
* No previously treatment of oral ulcers with topical steroids, vitamins, antibiotics, antihistamines, oral retinoids, or immunomodulatory agents within three months prior to entering the study;
* No non-steroidal anti-inflammatory drugs or mouthwash administrations for the treatment of the ulcer within 72 hours before entering the study.
* Pregnants or breastfeeding patients.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-02-24 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 14 days
  Pain intensity, measured using the VAS (Visual Analogue Scale), consisting of a 10 cm line, where 0 indicates no pain and 10 indicates intense pain.
Ulcers Dimensions | 14 days
  Size of each ulcer measured through a sheet of clear plastic will be applied directly to the ulcer by tracing the circumference of the ulcer and then placed on a graph paper and the number of mm2 units included within the drawn area will be counted.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Antonio Scarano Antonio Scarano, MD DDS, Study Director — Department of Innovative Technology in Medicine and Dentistry
Locations (1):
- University of Chieti- Department of Innovative Technology in Medicine and Dentistry, Chieti, Abruzzo, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/61/NCT07121361/Prot_SAP_000.pdf